CLINICAL TRIAL: NCT06052930
Title: Immersive Virtual Reality for the Non-pharmacological Management of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Neurológico Sénior (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNS-11-2022
Record Dates: First submitted 2023-08-14; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: Immersive virtual reality; Neurorehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): 12 consecutive weeks of physiotherapy + training with the IVR
  Interventions: Device: HTC Vive™ Pro
- Active control group (Active Comparator): 6 consecutive weeks of physiotherapy only, followed by 6 consecutive weeks of physiotherapy + training with the IVR
  Interventions: Device: HTC Vive™ Pro

INTERVENTIONS:
Device: HTC Vive™ Pro — A commercially available head-mounted display. Each VR session has approximately 20 minutes, performed 3 times per week.
  Both groups maintain similar PD specialized physiotherapy sessions throughout the duration of the study (3 times per week, 60 minutes per session).

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility, safety and efficacy of an immersive virtual reality (IVR) exergaming using a head-mounted display in Parkinson's disease symptomatic control.

This is a parallel-group, single-blinded, randomized controlled trial. The intervention group perform 12 weeks of physiotherapy and IVR, whereas the control group have 6 weeks of physiotherapy only, followed by 6 weeks of physiotherapy and IVR. The primary outcome is the symptomatic effect of the intervention as measured by the change from baseline in Time Up and Go (TUG) test with cognitive dual-task (TUG cognitive).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Parkinson's disease according to MDS criteria;
* Hoehn and Yahr stages between I-III (MED ON);
* Ability to perform the Time Up and Go test in normal pace and without assistance, in less than 11,5 seconds in ON state;
* Stable medication for the past 1 month;
* Ability to communicate with the investigator, to understand and comply with the requirements of the study;
* Able to provide written informed consent to participate in the study.

Exclusion Criteria:

* Postural instability or freezing of gait in MED ON representing an increased risk of fall, according to the best clinical judgement;
* A Montreal Cognitive Assessment (MoCA) score < 21;
* Presence of severe visual loss that could interfere with the ability to see the VR simulation as well as vertigo, epilepsy and psychosis;
* Unstable medical condition, including cardiovascular, pulmonary or musculoskeletal, that according to the clinician's judgment affect patients' ability to participate in the study;
* Inability to correctly respond to the assessment protocol according to the clinician's judgment or lack of support from caregiver for this effect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-19 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2023-08-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 6-week in TUG cognitive test | 6 week
  Change from baseline to 6-week in TUG cognitive test

SECONDARY OUTCOMES:
Change from baseline to each evaluation time point in TUG and TUG with motor and cognitive dual-tasking | 6, 12 and 16 weeks
  Difference between groups in change from baseline to each evaluation time point in TUG and TUG with motor and cognitive dual-tasking
Change from baseline to each evaluation time point in MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 6, 12 and 16 weeks
  Difference between groups in change from baseline to each evaluation time point in MDS-UPDRS
Change from baseline to each evaluation time point in mini-Balance Evaluation Systems Test (mini-BEST test) | 6, 12 and 16 weeks
  Difference between groups in change from baseline to each evaluation time point in mini-BEST test
Change from baseline to each evaluation time point in Montreal Cognitive Assessment (MoCA) | 6, 12 and 16 weeks
  Difference between groups in change from baseline to each evaluation time point in MoCA
Change from baseline to each evaluation time point in Stroop test | 6, 12 and 16 weeks
  Difference between groups in change from baseline to each evaluation time point in Stroop test
Change from baseline to each evaluation time point in Visual Object and Space Perception (VOSP) Battery (cube and fragmented letters) | 6, 12 and 16 weeks
  Difference between groups in change from baseline to each evaluation time point in VOSP-cube analysis and VOSP-fragmented letters
Change from baseline to each evaluation time point in Parkinson's Disease Questionnaire-39 items (PDQ-39) | 6, 12 and 16 weeks
  Difference between groups in change from baseline to each evaluation time point in PDQ-39 score
Change from baseline to each evaluation time point in Schwab and England (S&E) scale | 6, 12 and 16 weeks
  Difference between groups in change from baseline to each evaluation time point in S&E scale
Change from baseline to each evaluation time point in Clinical and Patient Global Impression of severity | 6, 12 and 16 weeks
  Difference between groups in change from baseline to each evaluation time point in Clinical and Patient Global Impression of severity
Change from baseline to each evaluation time point in BMI | 6, 12 and 16 weeks
  Difference between groups in change from baseline to each evaluation time point in BMI
Occurrence of adverse events | 16 weeks
  Difference between groups in patient's safety
Occurrence of cybersickness using the Simulator Sickness Questionnaire (SSQ) | 16 weeks
  Difference between groups in SSQ
Patients' consideration on system usability using the System Usability Scale (SUS) | 1, 6, 12 and 16 weeks
  SUS after the 1st week using the IVR system and at each evaluation time point
Patients' Borg perceived exertion | 16 weeks
  Difference between groups in perceived exertion
Likert scale on patients' satisfaction using the virtual reality system | 12 weeks
  Difference between groups in patients' satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Ferreira, MD, PhD, Study Director — CNS-Campus Neurologico
Locations (1):
- CNS-Campus Neurológico, Lisbon, Portugal